CLINICAL TRIAL: NCT06884319
Title: Diagnostic Accuracy of the Optic Nerve Deformability Index and Optic Nerve Sheath Diameter as a Noninvasive Predictor of Intracranial Pressure
Status: Active, not recruiting | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ghada Mohamed Ali Ibrahim El sokkary, Assistant lecturer, Benha University
Other Study IDs: MD 15_2_2025
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Increase Intra Cranial Pressure; Traumatic Brain Injury
Keywords: Optic nerve sheat diameter; Deformability index; Increase intra cranial pressure
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The study will be carried out on 50 patients, dichotomized into high and normal ICP groups, and we will assess both ONSD and DI in all patients.

DETAILED DESCRIPTION:
Operational Design:

Preparation:

Awake and alert patients should be briefed on the procedure. Obtunded, intubated, or heavily sedated patients should undergo a basic eye evaluation for signs and symptoms of globe rupture or hyphema. If there is evidence of globe rupture-including visible conjunctival or scleral defects, severe chemosis, 360-degree conjunctival hemorrhage, hypotony, or total hyphema-the procedure should be aborted to avoid further herniation of intraocular contents, and an ophthalmologist should be consulted. The patient's position should be determined by comfort and ease of examination, but the procedure will typically be performed in a supine to 30-degree "head-up" position. Although theoretical concerns may exist regarding changes in ICP and optic nerve sheath diameter (ONSD) relative to patient position and ventilator settings, these changes do not appear to manifest in vivo.

Methods:

1. Optic Nerve Sheath Diameter (ONSD) Assessment:

   After applying a generous amount of ultrasound gel, the high-frequency ultrasound linear transducer should be placed over the eye in the transverse plane. The sonographer's hand should rest on a non-compressible surface (such as the patient's nose, midface, or forehead) to avoid direct pressure on the globe, discomfort, and anatomical distortion. Small movements in the nasal and temporal directions, followed by caudal and cephalic adjustments, should be performed to capture the optic nerve sheath in the same plane as the lens, thus avoiding an oblique image. Once the anechoic streak posterior to the optic disc is visualized, the image should be captured, and measurements can be taken from the saved image. The optic nerve is relatively cylindrical and symmetrical, which theoretically makes a single view acceptable for measurement.

   Point of Measurement for ONSD:

   Three millimeters from the optic disc, posterior to the globe, corresponds to the bulbous (widest) portion of the optic nerve and is the site of maximum pressure changes within the nerve. For each optic nerve, two measurements are made-one in the sagittal plane and the other in the transverse plane (by rotating the probe clockwise). The mean value obtained for both eyes is retained as the final ONSD value.
2. Deformability Index (DI) Assessment:

The deformability index (DI) of the optic nerve sheath (ONS) can be assessed using ultrasound to evaluate changes in intracranial pressure (ICP). This technique involves observing how the optic nerve sheath diameter (ONSD) changes in response to pressure or dynamic forces. It is based on the hypothesis that raised ICP leads to increased stiffness of the ONS complex due to the accumulation of CSF, thereby reducing its ability to deform under cardiovascular pulsation. The Deformability Index (DI) was calculated according to the method described by Padayachy et al. (2016), which estimates the magnitude of motion (D1 and D2) in the lateral direction on both sides of the ONS over the cardiac cycle. This dimensionless parameter quantifies the deformation of the nerve sheath complex according to the formula.

The method depends on the manual initialization of two points. To reduce operator dependency, the initialization was standardized by drawing a central, straight line through the optic nerve axis, with perpendicular measurements of the DI at predefined depths from the sclera. Results at 3.0 mm, 3.5 mm, and 4.0 mm depths will be calculated, and the average values will be used in further analysis. For patients in whom ultrasound acquisitions from both eyes were obtained, the average of the left and right eyes was calculated and used as the DI value in further analysis.

Normal DI: Indicates a compliant optic nerve sheath, suggesting normal ICP. Reduced DI: Suggests decreased compliance of the optic nerve sheath, typically seen in elevated ICP due to rigid structures limiting deformation.

Administrative and Ethical Design:

Approval from the Research Ethics Committee of Benha Faculty of Medicine will be obtained. Informed written consent will be obtained from all patients or their first-degree relatives before participation. The consent will include information about the aim of the study, study design, site, timing, subject details, methods, and confidentiality.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 65 years
* increased ICP (e.g., TBI, sub arachnoid hemorrhage, intracranial hemorrhage)
* a Glasgow Coma scale=3-12 and requiring ICP monitoring via invasive methods (e.g. extra ventricular drain, lumber drain)

Exclusion Criteria:

* chronic hydrocephalus
* extensive local orbit trauma
* a pre-existing ocular disease affecting the optic nerve and/or orbital cavity
* hyperthyroidism with exophthalmia
* facial trauma affecting the orbits and/or eyeballs
* optic nerve trauma
* signs of critically raised ICP, needing urgent surgery.
* hemodynamically unstable between ONSD acquisition and ICP measurement.
* receiving medication that would decrease ICP between ultrasound imaging and ICP measurement, i.e. mannitol, hypertonic saline or steroids.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be carried out on 50 patients, dichotomized into high and normal ICP groups and we will assess both ONSD and DI in all patients.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Detect increase intra cranial pressure | 1 week
  By detection of increase intra cranial pressure early and rabid by Ultrasound we can treat early and avoid side effects of invasive measures

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Mostafa Abd El-hamed, Professor, Study Director — Benha University
Locations (1):
- Benha university hospital, Banhā, Egypt